CLINICAL TRIAL: NCT06212817
Title: FiberUP in Clinical Practice: Increasing Preoperative Dietary Fiber Intake in Colorectal Cancer Patients.
Brief Title: Dietary Fiber Before Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Gelderse Vallei Hospital (Other); VLAG Graduate School (Unknown); Alliance TU/e, WUR, UU, UMC Utrecht (EWUU) (Unknown); Nutrition & Healthcare Alliance (Unknown); WholeFiber BV (Unknown); Wageningen Food and Biobased Research (WFBR) (Unknown); Meander Medical Center (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Dieuwertje Kok, Associate Professor, PhD, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-16470; NL84650.091.23 (Other: METC Oost-Nederland)
Record Dates: First submitted 2023-12-05; First posted 2024-01-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: Dietary fiber; Postoperative complications; Surgery; Gut microbiota; Colorectal cancer; Prehabilitation
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with three parallel arms consisting of two intervention arms and one control arm. Multicenter study conducted in collaboration with three participating hospitals, including Hospital Gelderse Vallei (Ede), Meander Medical Center (Amersfoort), and Rijnstate Hospital (Arnhem)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fibre-UP tool: digital, personalized dietary advice to increase dietary fiber intake (Experimental): Subjects will receive personalized dietary advice (PDA) based on their habitual food pattern (as assessed using a food frequency questionnaire) and preferences. Based on a previously developed algorithm, the PDA provides fiber-rich alternatives for currently used low-fiber products, close to subjects' current eating behavior, to help increase dietary fiber intake. This PDA will be provided using an online web-portal.
  Interventions: Other: Dietary intervention
- Vegetable product (dried chicory root) to increase dietary fiber intake (Experimental): Subjects will consume 2 sachets with each 7.5 g of dried cubes of chicory root, which equals a total of 12.3 g of dietary fiber per day. Subjects can choose when and how they consume the vegetable product, for example sprinkle it over their meal, or include in existing recipes.
  Interventions: Other: Dietary intervention
- Control (No Intervention): Subjects will follow their habitual diet during the preoperative period.

INTERVENTIONS:
Other: Dietary intervention — Increase dietary fiber intake
  Arms: Fibre-UP tool: digital, personalized dietary advice to increase dietary fiber intake; Vegetable product (dried chicory root) to increase dietary fiber intake

SUMMARY:
The aim of this randomized controlled trial is to investigate the feasibility of increasing preoperative dietary fiber intake in individuals with colorectal cancer who will undergo surgery. This will be done using 1) digital personalized dietary advice or 2) a dried vegetable product compared to 3) habitual diet (control).

DETAILED DESCRIPTION:
Rationale: Postoperative complications, affecting up to 50% of the patients with colorectal cancer (CRC) undergoing surgery, are associated with impaired quality of life and higher mortality rates. The investigators have previously shown an association between a higher preoperative dietary fiber intake and a lower risk of postoperative complications. Before large interventions aiming to evaluate potential causal relationships between dietary fiber and postoperative complications can be implemented, feasibility of increasing dietary fiber intake before CRC surgery needs to be explored.

Objective: To investigate the feasibility of increasing preoperative dietary fiber intake in CRC patients undergoing surgery via 1) personalized dietary advice (Vezel-UP tool), or 2) vegetable product containing natural fibers compared to 3) habitual diet (control group). Secondary objectives will be considered to generate preliminary (biological) data to support the design of a future large-scale intervention studies.

Study design: A randomized controlled trial with three groups: 1) Vezel-UP group, 2) vegetable product group, and 3) control group. The intervention period equals the time between diagnosis and surgery, which is on average ~4 weeks but will vary between individual patients depending on their characteristics (e.g., physical condition and tumor location) and waiting list.

Study population: 54 CRC patients who will undergo elective tumor resection.

Main study parameters/endpoints: The primary outcome is the change in dietary fiber intake, which is assessed via two 24hr dietary recalls at baseline and during and after the intervention. Secondary parameters are stool pattern, gastrointestinal symptoms, quality of life, fecal microbiota composition, fecal and plasma microbial metabolites levels (i.e., SCFA and indoles), and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Being diagnosed with CRC and planned to undergo elective CRC resection;

Exclusion Criteria:

* Previously have had a large abdominal resection, excluding appendectomy and cholecystectomy;
* Diagnosed with Crohn's disease, Ulcerative Colitis, Celiac Disease;
* Currently having a stoma;
* Known allergic reactions to plants from the Asteraceae (Compositae) family (e.g., lettuce, daisies, sunflowers, artichokes, sage, tarragon, chamomile, chicory etc.);
* Currently following a strict diet and unwilling or unable to change (e.g., gluten free or ketogenic diet);
* Currently using fiber supplements, prebiotics and/or probiotics and unwilling to stop using these for the duration of the intervention;
* Having a habitual dietary fiber intake >30 g/day for women and >40 g/day for men, measured with a food frequency questionnaire;
* Dementia or other cognitive disabilities that makes it impossible to fill out questionnaires correctly;
* Illiteracy (inability to read and understand Dutch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Dietary fiber intake | 3 time points: T0 (at baseline), T1 (after 2 weeks of intervention), and T2 (at the end of intervention period, on average after 4 weeks).
  Change in dietary fiber intake is assessed via two 24hr dietary recalls.

SECONDARY OUTCOMES:
Stool pattern | 3 time points: T0 (at baseline), T1 (after 2 weeks of intervention), and T2 (at the end of intervention period, on average after 4 weeks).
  Change in stool frequency per week and average stool consistency per week assessed using the Bristol Stool Chart.
Gastrointestinal symptoms | 3 time points: T0 (at baseline), T1 (after 2 weeks of intervention), and T2 (at the end of intervention period, on average after 4 weeks).
  Change in gastrointestinal symptoms measured with the Gastrointestinal Symptom Rating Scale (GSRS). Higher scores mean a worse outcome.
Health-related quality of life | 3 time points: T0 (at baseline), T1 (after 2 weeks of intervention), and T2 (at the end of intervention period, on average after 4 weeks).
  Change in quality of life measured with the European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (EORTC QLQ-C30 & CR29). Global and functional health-related quality of life will be calculated, for which higher scores indicate better quality of life. Also symptom scales will be calculated, for which higher scores indicate higher presence or severity of a symptom.
Fecal gut microbiota composition | 3 time points: T0 (at baseline), T1 (after 2 weeks of intervention), and T2 (at the end of intervention period, on average after 4 weeks).
  Measured using 16S rRNA amplicon sequencing in fecal samples.
Fecal microbial metabolite levels | 3 time points: T0 (at baseline), T1 (after 2 weeks of intervention), and T2 (at the end of intervention period, on average after 4 weeks).
  Change in SCFA and indole concentrations determined by GC-MS/MS and LC-MS/MS in fecal samples.
Plasma microbial metabolite levels | 2 time points: T0 (at baseline) and T2 (at the end of intervention period, on average after 4 weeks).
  Change in SCFA and indole concentrations will be determined by GC-MS/MS and LC-MS/MS in blood samples.
Length of hospital stay | From date of surgery until date of hospital discharge, assessed up to 90 days after surgery.
  Time between surgery and hospital discharge in number of days based on data from medical records.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Rijnstate, Arnhem, Gelderland
  - Ziekenhuis Gelderse Vallei, Ede, Gelderland
  - Meander Medisch Centrum, Amersfoort, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kok DE, Arron MNN, Huibregtse T, Kruyt FM, Bac DJ, van Halteren HK, Kouwenhoven EA, Wesselink E, Winkels RM, van Zutphen M, van Duijnhoven FJB, de Wilt JHW, Kampman E. Association of Habitual Preoperative Dietary Fiber Intake With Complications After Colorectal Cancer Surgery. JAMA Surg. 2021 Jun 16;156(9):1-10. doi: 10.1001/jamasurg.2021.2311. Online ahead of print. PMID 34132738
- [Background] Rijnaarts I, de Roos NM, Wang T, Zoetendal EG, Top J, Timmer M, Bouwman EP, Hogenelst K, Witteman B, de Wit N. Increasing dietary fibre intake in healthy adults using personalised dietary advice compared with general advice: a single-blind randomised controlled trial. Public Health Nutr. 2021 Apr;24(5):1117-1128. doi: 10.1017/S1368980020002980. Epub 2020 Sep 18. PMID 32943128
- [Background] Rijnaarts I, de Roos NM, Wang T, Zoetendal EG, Top J, Timmer M, Hogenelst K, Bouwman EP, Witteman B, de Wit N. A high-fibre personalised dietary advice given via a web tool reduces constipation complaints in adults. J Nutr Sci. 2022 Apr 28;11:e31. doi: 10.1017/jns.2022.27. eCollection 2022. PMID 35573462
- [Background] Puhlmann ML, Jokela R, van Dongen KCW, Bui TPN, van Hangelbroek RWJ, Smidt H, de Vos WM, Feskens EJM. Dried chicory root improves bowel function, benefits intestinal microbial trophic chains and increases faecal and circulating short chain fatty acids in subjects at risk for type 2 diabetes. Gut Microbiome (Camb). 2022 Apr 28;3:e4. doi: 10.1017/gmb.2022.4. eCollection 2022. PMID 39295776